CLINICAL TRIAL: NCT06320054
Title: Preventing Common Obstetric Complications Through an Immersive, Medically Tailored Meal Program
Brief Title: Preventing Obstetric Complications With Dietary Intervention
Acronym: PLATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Advancing a Healthier Wisconsin Endowment (Unknown); Food for Health, Inc. (Unknown)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00049771
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes; Gestational Hypertension; High Risk Pregnancy; Preeclampsia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Prenatal Care (No Intervention): Standard Prenatal Care, biometric screenings, and surveys (baseline, 4-12 weeks postpartum).
- Maternal Health Management Program (Experimental): Program participants will receive 10 fresh, local meals each week, delivered to their homes, health coaching including cooking and physical activity, biometrics screenings, and educational support to enable sustainable lifestyle change.
  Interventions: Behavioral: Maternal Health Management Program

INTERVENTIONS:
Behavioral: Maternal Health Management Program — Program participants will receive 10 fresh, local meals each week, delivered to their homes, health coaching including cooking and physical activity, biometrics screenings, and educational support to enable sustainable lifestyle change.
  Arms: Maternal Health Management Program

SUMMARY:
The goal of this study is to learn whether access to healthy and fresh food, health coaching, and nutrition support intervention can reduce adverse birth outcomes in pregnant women. The main questions it aims to answer are:

* Does access to healthy and fresh food, health coaching and nutrition support reduce the risk of gestational diabetes or preeclampsia and ultimately improve health outcomes for mothers and their newborns?
* Are participants able to successfully utilize the health program? Are participants satisfied and self-equipped to apply the teachings of the program within their lives following their participation in the study? Participants will be randomly assigned to one of two groups.

Participants in the standard of care will be asked to:

* Complete surveys
* Biometric screenings

Participants in the intervention group will be asked to:

* Complete surveys
* Biometric screenings
* Participate in weekly personal health coaching
* Receive and consume provided weekly meals.

Researchers will compare the standard of care to those who receive the intervention to see the impact of the intervention on clinical outcomes including: gestational weight gain, blood pressure, diagnosis of gestational diabetes, diagnosis of gestational hypertension or preeclampsia, and gestational age at birth.

ELIGIBILITY:
Inclusion criteria:

1. Age at enrollment ≥ 18 years of age
2. Receiving prenatal care at Froedtert
3. ≤ 16 weeks and 6 days of gestation
4. At risk of preeclampsia, defined as being eligible for low dose aspirin treatment AND/OR at risk for gestational diabetes defined as having a history of gestational diabetes, OR previously given birth to an infant weighing ≥ 4000 g, OR has a diagnosis of PCOS
5. Pre-pregnancy Body Mass Index ≥ 25 kg/m^2
6. Resides in Milwaukee County at time of consent
7. Low socio-economic status (<200% of FPL defined as receiving Medicaid)
8. Able to read and communicate in English
9. Has access to a smart device/computer with reliable internet connection
10. Has access to a working refrigerator
11. Viable singleton pregnancy

Exclusion criteria:

1. Diagnosed with Type I or Type II Diabetes or Hemoglobin A1C ≥ 6.5%
2. Diagnosed with End Stage Renal Disease
3. Use of weight-increasing psychotropic agents
4. Active inflammatory bowel disease, or history of bowel resection or malabsorptive syndrome, or history of bariatric surgery
5. Significant food allergies, preferences or dietary requirements that would interfere with diet adherence
6. Multifetal gestation
7. Active substance use that would preclude program adherence
8. Chronic use of oral corticosteroids
9. Unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  gestational weight gain (BMI early pregnancy in comparison to BMI at delivery)
Clinical Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  blood pressure (Compared to early pregnancy, intrapartum, postpartum
Clinical Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  Diagnosis of gestational diabetes
Clinical Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  Diagnosis of preeclampsia or gestational hypertension
Clinical Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  Gestational age at birth (Weeks and Days)

SECONDARY OUTCOMES:
Patient Reported Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  program utilization (measured by percentage of weekly coaching attended and number of meals consumed)
Patient Reported Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  participant satisfaction and retention (measured by end of study evaluation)
Patient Reported Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  self-efficacy skills with meals preparation (as measured by nutrition survey)
Patient Reported Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  physical activity planning (as measured by physical activity survey)
Patient Reported Outcomes | End of Pregnancy up to 8 weeks postpartum (+/- 2 weeks)
  Self-Efficacy (as measure by Self-Efficacy survey)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedert & The Medical College of Wiscosin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided